CLINICAL TRIAL: NCT07202416
Title: Comparison of Erector Spinae Plane Block and Intrathecal Morphine for Assessements of Quality of Recovery After Caesarean Section: a Randomized Controlled Trial
Brief Title: ESPB vs Intrathecal Morphine for Assessements of Quality of Recovery After Cesarean Section
Acronym: BELLMERE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AUSL Romagna Rimini (Other)
Responsible Party: Principal Investigator, Domenico Pietro Santonastaso, MD, AUSL Romagna Rimini
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2223/2025 I.5/33
Record Dates: First submitted 2025-07-15; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Cesarean Section; Post Operative Pain
Keywords: Cesarean Section; Erector Spinae plane block; Quality of recovery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (Experimental): Patients in this group will receive an ultrasound-guided bilateral Erector Spinae Plane Block at the end of cesarean section, in addition to standard spinal anesthesia without intrathecal morphine.
  Interventions: Procedure: Erector spinae plane block
- Intrathecal MorphineITM (Active Comparator): Patients in this group will receive a standard dose of intrathecal morphine during spinal anesthesia for cesarean section. No additional fascial plane block will be performed.
  Interventions: Procedure: Intrathecal morphine

INTERVENTIONS:
Procedure: Erector spinae plane block — Ultrasound-guided Erector Spinae Plane Block performed at the T9 level with 0,375%, ropivacaine 20 mL administered bilaterally at the end of surgery for postoperative analgesia following cesarean section.
  Other Names: ESPB
  Arms: Erector Spinae Plane Block
Procedure: Intrathecal morphine — Intrathecal administration of 100 mcg of morphine in combination with a local anesthetic was performed at the time of spinal anesthesia for cesarean section.
  Other Names: ITM
  Arms: Intrathecal MorphineITM

SUMMARY:
Cesarean section is a surgical procedure that involves significant pain, which is managed through a multimodal pharmacological approach.The primary objective of the study is to evaluate the quality of hospitalization after cesarean section using the QRo11 questionnaire in patients treated with a postoperative Erector Spinae Plane Block compared to those treated with intrathecal morphine.

DETAILED DESCRIPTION:
Cesarean section is one of the most common surgical procedures worldwide and is associated with significant postoperative pain. Effective pain control is crucial to enhance maternal recovery, improve mobilization, support breastfeeding, and reduce hospital stay. Traditionally, intrathecal morphine has been widely used as part of a multimodal analgesic regimen. However, its use may be limited by opioid-related side effects such as nausea, vomiting, pruritus, and respiratory depression.

Regional anesthesia techniques targeting the thoracic paravertebral space have recently been introduced to improve postoperative pain control while reducing opioid consumption. The Erector Spinae Plane (ESP) Block is a relatively simple and safe fascial plane block that has shown promising results in different surgical settings, including obstetric procedures.

The primary aim of this prospective study is to evaluate the quality of recovery after cesarean section using the validated Quality of Recovery-11 (QoR-11) questionnaire. Patients will be allocated to receive either a postoperative ESP block or intrathecal morphine as part of their analgesic protocol.

Secondary endpoints include postoperative pain scores, opioid consumption, incidence of opioid-related side effects, time to mobilization, breastfeeding outcomes, and duration of hospital stay.

This study will provide new evidence on the role of the ESP block in cesarean section and may contribute to optimizing multimodal analgesia strategies for mothers undergoing this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult women aged 18-45 years
* ASA physical status II-III
* Full-term singleton pregnancy scheduled for elective cesarean section under spinal anesthesia

Exclusion Criteria:

* ASA ≥ IV
* Coagulation disorders
* Emergency surgery
* Preoperative infection (including infection at the ESPB puncture site)
* Any contraindication to neuraxial analgesia
* History of chronic pain
* Use of opioids
* Allergy to local anesthetics
* Hypersensitivity to any drug used in the study
* Inability to understand or use verbal pain assessment scales
* Refusal to participate in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
QoR-11 questionnaire score | day 1 after surgery
  Assessment of QoR-11 questionnaire score

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) pain scores | 4, 6, 8, 12, and 24 hours after cesarean section
  Assessment of Numerical Rating Scale (NRS) pain scores both at rest and during movement. NRS 0-10. 0 mean a better outcome, 10 mean a worse outcome.
rescue dose | day 1 after surgery
  Time to first rescue dose (interval between the block or intrathecal morphine administration and the first request for opioid analgesia).
complications | day 1 after surgery
  Assessment of adverse events such as sedation, nausea, and other complications
breastfeeding latch | day 1 after surgery
  Time from birth to first breastfeeding latch

CONTACTS AND LOCATIONS:
Overall Officials: Domenico P Santonastaso, MD, Principal Investigator — AUSL Romagna - M. Bufalini Hospital
Locations (1):
- AUSL Romagna - Ospedale M.Bufalini, Cesena, Forlì, Italy